CLINICAL TRIAL: NCT06026215
Title: Assessing the Effects of Mechanical Unloading on Tissue and Immunologic Characteristics Indictive of Cardiac Repair
Brief Title: Assessing the Effects of Mechanical Unloading on Repair Version-1
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2015CD001; 139009 (Other: IRAS ID)
Record Dates: First submitted 2023-08-04; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Heart Failure; Transplant; Failure, Heart
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Heart failure patients requiring ventricular assist device implantation will be included into group 1.
- Group 2: Heart transplant recipients requiring early extracorporeal membrane oxygenation will be recruited into group 2.
- Group 3: Heart transplant recipients who have not previously received a VAD will be recruited into group 3.

SUMMARY:
The mechanism by which heart failure initiates and progresses and the mechanisms of heart repair remain unclear.

The left ventricular assist device (LVAD) is a therapy to stabilise patients while they await their transplant. The LVAD helps pump blood around the body, giving the heart an opportunity to recover. During surgery, the apical core tissue is routinely removed to allow the implantation of the device (this tissue is normally discarded). Some patients demonstrate cardiac recovery, allowing the device to be removed without later needing a transplant. As part of the LVAD removal procedure, the section around the device might need to be removed (this tissue is normally discarded). To further understand the cellular and molecular mechanisms by which the heart is repaired, the investigators wish to utilise this surplus tissue for research purposes. The collection of this tissue is part of routine treatment and does not represent additional risk for the patient for research purposes. Some patients might still require a transplant following VAD treatment. The native heart is removed from these patients (routinely discarded) and replaced by a donor heart. The investigators wish to utilise this discarded tissue for research purposes, so that the investigators can identify the cellular and molecular factors involved in cardiac repair and which distinguish responsive and non-responsive patients. Heart transplant recipients who require extracorporeal membrane oxygenation will have an additional heart biopsy sample taken for research purposes when performed as part of routine clinical practice. There is no additional risk to the patient for research purposes. Heart failure patients scheduled for transplantation (who have not received a VAD) will be recruited prior to transplantation and their native heart retained for research purposes. An additional peripheral blood sample will be collected from all patients for research purposes when performed for routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to provide informed consent; informed consent may be provided retrospectively if this cannot be provided pre-surgery.
* Patients must be aged between 18--70 years of age.
* Patients who have been clinically diagnosed with chronic heart failure and require mechanical unloading using a left ventricular assist device.
* Patients who have received a heart transplant but require extracorporeal membrane oxygenation.

Exclusion Criteria:

* Patients under 18 or over 70 years of age.
* Patients unable to provide informed consent.
* Patients who are prisoners.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic heart failure and require mechanical unloading using a left ventricular assist device.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in protein expression within the tissue during clinical repair. | through study completion - 4 years
  Relate small changes in protein expression within the heart tissue to clinical parameters indicative of function. Additionally, the investigators aim to extend our understanding of the mechanisms underpinning heart failure by identifying the factors responsible for either preventing repair or promoting expedited disease progression.